CLINICAL TRIAL: NCT00653588
Title: A 26-Week, Double Blind, Randomised, Multi-Centre, Phase IIIb, Parallel Group Study to Compare the Efficacy and Safety of Rosuvastatin (40 mg) With Atorvastatin (80 mg) in Subjects With Hypercholesterolaemia and Coronary Heart Disease or CHD Risk Equivalents
Brief Title: Polaris - Crestor 40 mg vs Atorvastatin 80 mg for 26 Weeks
Acronym: POLARIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522IL/0106; D3569C00005
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: Cholesterol; low density lipoproteins; Hypercholesterolemia; Coronary Heart Disease; Rosuvastatin; Crestor; Atorvastatin; Lipitor
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): rosuvastatin (40 mg)
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): atorvastatin (80 mg)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 40mg
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin — 80mg
  Other Names: Lipitor
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of 8 weeks of treatment with Rosuvastatin with 8 weeks of treatment with Atorvastatin on low density lipoprotein cholesterol level in subjects with hypercholesterolemia and coronary heart disease (CHD) or at high risk of CHD..

ELIGIBILITY:
Inclusion Criteria:

* A history of CHD or clinical evidence of atherosclerosis or multiple risk factors that confer a high risk as defined in the protocol.
* Fasting LDL-C concentrations at Visit 1 as defined in the protocol.

Exclusion Criteria:

* History of statin induced serious side effects, or serious hypersensitivity reaction to other statins.
* Subjects considered to be unstable by the investigator after the following events: a myocardial infarction (heart attack), unstable angina, myocardial revascularisation or another revascularisation procedure or a transient ischaemic attack (TIA) or stroke.
* Severe congestive cardiac failure (as defined by the protocol - Appendix I).
* Subjects awaiting a planned myocardial revascularisation prior to starting the study (i.e. planned prior to visit 1).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of rosuvastatin with atorvastatin by assessing the percentage change from baseline to week 8 in LDL-C concentrations in subjects with hypercholesterolaemia and CHD or CHD risk equivalents.

SECONDARY OUTCOMES:
To compare the efficacy of rosuvastatin with atorvastatin in modifying other lipids and lipoproteins at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lawrence Leiter, Principal Investigator — St Michaels hospital, Canada